CLINICAL TRIAL: NCT01902914
Title: Effectiveness of NECTEC Model, Body-worn, Digital Hearing Aids and Cost of Screening and Hearing Aids Service in Elders
Brief Title: Effectiveness of P02 Digital Hearing Aids
Acronym: P02
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kwanchanok Yimtae, M.D., Assoc. Prof. Kwanchanok Yimtae, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HE551268
Record Dates: First submitted 2012-10-01; First posted 2013-07-18 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hearing Loss, Bilateral; Sensorineural Hearing Loss
Keywords: hearing aids; hearing disability; community; hearing aids service
MeSH Terms: conditions — Hearing Loss, Bilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hearing Aids, Model P02 (Experimental): A body-worn, local made, digital hearing aids Hearing Aids evaluation
  Interventions: Procedure: Hearing Aids Evaluation
- Other hearing aids (Active Comparator): Other Hearing Aids, Hearing Aids Evaluation
  Interventions: Procedure: Hearing Aids Evaluation

INTERVENTIONS:
Procedure: Hearing Aids Evaluation — Functional Gain Sound field Speech Audiometry
  Other Names: Functional Gain

SUMMARY:
To test the effectiveness of body-worn, digital hearing aids, model 02 which is developed by the National Electronics and Computer Technology Center, Thailand.

DETAILED DESCRIPTION:
Hearing aids distribution and service system are limited accessed in hearing disabled people in developing countries. The local-made, body-worn, digital hearing aids is developed by the National Electronics and Computer Technology Center, Thailand. The effectiveness of this model will be compares with other standard body-worn, hearing aids in community elders. The functional gain, quality of sound, customers' satisfaction, and quality of life (EQ-5D, HHIE, HUI-3, IOI-HA) are main outcomes.The cost of Screening and hearing aids will be also investigated. The validity and reliability of several tools used such as the Thai-Hearing Handicap Inventory for elderly (HHIE) questionnaire, Music Test, Thai-Five Minute Hearing Test, and Khon Kaen Hearing Aids Evaluation are also studied.

ELIGIBILITY:
Inclusion Criteria:

* older than 60 years
* bilateral sensorineural hearing loss
* PTA (0.5-2 KHz) of better ear > 40 DB but <75 dB
* no deformity of pinna and ear canal
* new or unexperienced hearing aids user
* can communicate with Thai or local language

Exclusion Criteria:

* speech discrimination <40%
* suspected of retrocochlear lesion

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
functional gain | Immediate after hearing aids fitting
  Different of hearing threshold between aids and un-aids

SECONDARY OUTCOMES:
Satisfaction | immediate after hearing aids fitting
  Sound quality satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kwanchanok Yimtae, MD, Principal Investigator — Khon Kaen University
Locations (1):
- Phu Wieng district, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Kasemsiri P, Yimtae K, Thanawirattananit P, Israsena P, Noymai A, Laohasiriwong S, Vatanasapt P, Siripaopradith P, Kingkaew P. Effectiveness of a programable body-worn digital hearing aid for older adults in a developing country: a randomized controlled trial with a cross-over design. BMC Geriatr. 2021 Jul 23;21(1):437. doi: 10.1186/s12877-021-02325-4. PMID 34301203